CLINICAL TRIAL: NCT05169216
Title: Effects of a Cognitive-Behavioral Therapy Intervention on the Rowers of the Junior Spain National Team
Brief Title: Cognitive-Behavioral Therapy on Junior Rowers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Raquel Leirós-Rodríguez, PhD. Principal Investigator, Universidad de León
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPAROW21
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Water Sports; Cognitive Behavioral Therapy; Psychological Techniques; Experience; Stress; Motivation
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-Behavioral Therapy Group (Experimental): A mental training program was carried out with the following objectives: (a) to learn to manage their level of activation; (b) to train their ability to concentrate; (c) to optimize their self-confidence; (d) to learn to compete by improving their racing routines; and (d) to integrate mental training into their day-to-day life.
  The athletes worked in small groups of four athletes. In addition, the days that the psychologist attended the concentration, he was also present in the training sessions, with the aim of giving them feedback on the strategies acquired. The psychologist was present in various phases throughout the concentration and there was also a constant online monitoring. Each week, a sheet of tasks to be executed and a diary were provided to verify compliance with the guidelines.
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — Each week, a sheet of tasks to be executed and a diary were provided to verify compliance with the guidelines:
  1. Week 0. Familiarization: Information gathering
  2. 1st week. Self-knowledge and concentration: To know sports psychology and mental training. Information on beliefs and expectations in sport.
  3. 2nd week: To integrate daily mental training.
  4. 3rd week. Trust: To consolidate concentration activation. To integrate and build confidence (in oneself and in the team).
  5. 4th week. Application to sports tactics: To apply concentration strategies to your sports practice. To know those strategies that provide the best results for each athlete.
  6. 5th and 6th weeks: To integrate the content already provided.
  7. 7th week. Link with the team: To strengthen the bond between team members.
  8. 8th week. Daily routines: To improve the daily routine prior to the competition.
  9. 9th and 10th weeks: To integrate the content already provided.

SUMMARY:
A quasi-experimental study was carried out with the complete team of the Spanish youth team of Rowing (n = 16). The setting where the intervention took place was during the concentration prior to the 2020 European Rowing Junior Championships. The final assessment was carried out the week before the championship (after finishing the 10th week of intervention). Psychological variables were assessed using the Psychological Characteristics Related to Sport Performance Questionnaire.

DETAILED DESCRIPTION:
A quasi-experimental study was carried out with the complete team of the Spanish youth team of Rowing (n = 16). The setting where the intervention took place was during the concentration prior to the 2020 European Rowing Junior Championships (held in Belgrade between September 25th and 27th). The athletes were concentrated without leaving their accommodation during the eleven weeks prior to the championship. A total of 27 rowers started the concentration, of whom 16 were eventually selected to participate in the championship.

A mental training program was carried out with the following objectives: (a) to learn to manage their level of activation; (b) to train their ability to concentrate; (c) to optimize their self-confidence; (d) to learn to compete by improving their racing routines; and (d) to integrate mental training into their day-to-day life.

The athletes worked in small groups of four athletes. In addition, the days that the psychologist attended the concentration, he was also present in the training sessions, with the aim of giving them feedback on the strategies acquired. The psychologist was present in various phases throughout the concentration and there was also a constant online monitoring. Each week, a sheet of tasks to be executed and a diary were provided to verify compliance with the guidelines.

The initial assessment was carried out on the second day of the concentration after the explanation of the intervention to be carried out. The final assessment was carried out the week before the championship (after finishing the 10th week of intervention).

Psychological variables were assessed using the Psychological Characteristics Related to Sport Performance Questionnaire (CPRD) (Gimeno, Buceta, & Perez-Llantada, 2007), based on the Psychological Skills Inventory for Sports (PSIS) (Mahoney, Gabriel, & Perkins, 1987). The questionnaire consists of 55 items graded in a 5-option Likert scale (from totally disagree to totally agree). It also includes a response option "I do not understand" to avoid missing answers. CPRD includes five subscales: Stress Control (SC), Influence of Performance Evaluation (IPE), Motivation (M), Team Cohesion (TC), and Mental Skills (MS), showing acceptable values of internal consistency for the total scale (α = 0.85) and for most of the subscales (αSC = 0.88; αIPE = 0.72; αM = 0.67; αTC = 0.78; αMS = 0.34) (Gimeno, & Pérez-Llanta, 2010).

In addition, the following study variables were taken into account: gender, age, years of experience in the rowing discipline and the position achieved on the podium in the 2020 European Championships.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Spanish youth team of Rowing

Exclusion Criteria:

* Not wanting to participate in the intervention.
* Not wanting to participate in the evaluation sessions.
* Failure to provide informed consent for participation by parents or guardians.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Psychological variables | The initial assessment: second day of the concentration. Final assessment: week before the championship (after finishing the 10th week of intervention
  Psychological variables were assessed using the Psychological Characteristics Related to Sport Performance Questionnaire (CPRD) based on the Psychological Skills Inventory for Sports (PSIS).

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias de la Salud, Ponferrada, Spain

IPD SHARING:
Plan to Share IPD: Yes
To publish a scientific article with the results obtained.